CLINICAL TRIAL: NCT00566865
Title: A Double-Blind, Placebo-Controlled Study to Assess the Effect of Gemfibrozil Co-Administration on the Pharmacokinetics and Pharmacodynamics of Mitiglinide in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study of Mitiglinide and Gemfibrozil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elixir Pharmaceuticals (Industry)
Responsible Party: Paul Martha, Chief Medial Officer, Elixir Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX-1510-CT-002
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gemfibrozil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): mitiglinide + gemfibrozil
  Interventions: Drug: gemfibrozil
- 1 (Placebo Comparator): mitiglinide + placebo for gemfibrozil
  Interventions: Drug: placebo for gemfibrozil

INTERVENTIONS:
Drug: placebo for gemfibrozil — mitiglinide + placebo for gemfibrozil 600 mg bid
  Arms: 1
Drug: gemfibrozil — Mitiglinide + 600 mg gemfibrozil bid
  Arms: 2

SUMMARY:
The primary objective of this study is to determine the extent of effect of gemfibrozil on the pharmacokinetics and pharmacodynamics of mitiglinide.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker
* Body mass index (BMI) of 19-28 kg/m2
* no relevant food allergies

Exclusion Criteria:

* any subject for whom gemfibrozil is contraindicated
* any subject with a history of hypoglycemia or who tend to get easily hypoglycemic
* clinically significant history of or current abnormality or disease of any organ system

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of mitiglinide | 3 days of treatment with gemfibrozil
pharmacodynamics of mitiglinide | 3 days of treatment with gemfibrozil

SECONDARY OUTCOMES:
safety and tolerance of mitiglinide when co-administered with 600 mg gemfibrozil | 3 days of treatment with gemfibrozil

CONTACTS AND LOCATIONS:
Overall Officials: Erin Nulf, RN, BSN, Study Director — Quintiles Phase I Services